CLINICAL TRIAL: NCT03887832
Title: Small Moments, Big Impact; Supporting Maternal Empathy by Adding Media to Child Health Services
Brief Title: Small Moments Big Impact (SMBI)
Acronym: SMBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-38334
Record Dates: First submitted 2019-03-21; First posted 2019-03-25 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Empathy
Keywords: child development; maternal empathy; digital media-based pediatric intervention; small moments, big impact (SMBI)
MeSH Terms: interventions — Infant Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SBSI intervention (Experimental): Mothers is this arm will download the SMBI intervention app onto their smartphone. They will be shown a video from the app and how to share videos with others. After hospital discharge, mothers will receive a weekly media package (video, associated prompt(s), and activity) via the SMBI for six months.
  Interventions: Other: SMBI digital app; Behavioral: media package; Other: standard newborn and infant care
- Infant standard of care (Active Comparator): Mothers in this arm will receive the standard of care for newborn and infants including education and a list of resources.
  Interventions: Other: standard newborn and infant care

INTERVENTIONS:
Other: SMBI digital app — Digital platform on the smartphone for the media package
  Arms: SBSI intervention
Behavioral: media package — The SMBI app contains a <1 minute video of a mother and baby or just mother, a reflection question about the video, a few questions about their mood and stress, and some prompts and suggestions on what to do if they have problems.
  Arms: SBSI intervention
Other: standard newborn and infant care — Recommended standard pediatric primary care will be provided for infants up to 6 months.

SUMMARY:
Empathy is defined as sensitivity to the needs of others.Maternal empathy, or a mother's sensitivity to the needs of her child, is critical for healthy child development ,Small Moments, Big Impact: Supporting Maternal Empathy by Adding Media to Child Health Services (SMBI) will develop and pilot a media-based pediatric primary care intervention that aims to answer two Big Questions: 1) Can media sent by pediatricians to mothers from low-income backgrounds promote empathy? 2) Is there a feasible and scalable approach? If successful, SMBI will result in: 1) increased maternal empathy; 2) new evidence and knowledge about an effective approach for supporting empathy in mothers from low-income backgrounds; 3) acceptability, feasibility of administering, and therefore potential for scalability through standard pediatric care; 4) increased support of maternal empathy as a core component of pediatric care; and 5) increased support by other stakeholders (including medical professionals, child health care facilities, and funders) to further explore, expand, and ultimately rollout the intervention

DETAILED DESCRIPTION:
This mixed methods research design will assess whether a digital media-based pediatric primary care intervention can increase empathy in mothers of newborns from low-income backgrounds compared to the current standard of care. During their newborns' stay in the nursery following recruitment, eligible mothers will be assigned to the intervention or comparison group. Mothers in the intervention group will download the SMBI smartphone app onto their phone and be trained by a research assistant (RA) on the functionality of the app. Mothers will be shown a video from the app, and shown how to share videos with others, to respond to prompts, and to rate the video. These activities represent what mothers are asked to do at home throughout the intervention. After departing the hospital, mothers in the intervention group will receive a media package (video, associated prompt/s, and activity) via the SMBI app every week for six months. Mothers will be asked to watch the videos, respond to the prompts, do the activities, and rate the value of videos via the SMBI app. Mothers will be encouraged to share questions and comments with the child's pediatrician and to share the videos with their support network. Mothers in the comparison group will receive the standard of care.

Mothers in both groups will be asked to complete a questionnaire at the end of recruitment and at 6 month visit and at the 6 month visit the investigators will also video tape and code a five minute play interaction. In addition, a focus group will be conducted with some mothers in the intervention group.

As of April 2020 in compliance with institutional COVID-19 policies all recruitment and interventions are being done without in-person contact.

ELIGIBILITY:
Inclusion Criteria:

* Adult mothers with a singleton baby born at term without any significant medical problems
* Mothers who plan to obtain pediatric care at BMC
* Mothers who are English speaking and reading
* Mothers who have a smartphone (data plan will be supplied if needed)

Exclusion Criteria:

-Mothers with substance abuse problems

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2019-08-29 (Actual); Primary Completion 2021-03-02 (Actual); Study Completion 2021-03-02 (Actual)

PRIMARY OUTCOMES:
Change in perspective-taking assessed with the Interpersonal Reactivity Index | baseline, 6 months
  The Interpersonal Reactivity Index (IRI) was designed to assess empathy, defined as "the reactions of one individual to the observed experiences of another." It has 28 items using 5-point scales (A = does not describe me well to E = describes me very well). It has 4 sub-scales: fantasy which assesses the extent to which individuals identify with fictional characters; perspective-taking which assesses the extent to which individuals spontaneously (try to) adopt others' points of view; empathetic concern which assesses the extent of individuals' "feelings of warmth, compassion, and concern for others."; and personal distress which assesses the extent of individuals "feelings of anxiety and discomfort" as a result of "another's negative experience." Each of the 4 sub-scales has 7 items and scores range from 28 to 140.
Change in empathetic concern assessed with the Interpersonal Reactivity Index | baseline, 6 months
  The Interpersonal Reactivity Index (IRI) was designed to assess empathy, defined as "the reactions of one individual to the observed experiences of another." It has 28 items using 5-point scales (A = does not describe me well to E = describes me very well). It has 4 sub-scales: fantasy which assesses the extent to which individuals identify with fictional characters; perspective-taking which assesses the extent to which individuals spontaneously (try to) adopt others' points of view; empathetic concern which assesses the extent of individuals' "feelings of warmth, compassion, and concern for others."; and personal distress which assesses the extent of individuals "feelings of anxiety and discomfort" as a result of "another's negative experience." Each of the 4 sub-scales has 7 items and scores range from 28 to 140.
Parent-infant interactions assessed with ORCE | 6 months
  Parent-infant videotaped interactions will be assessed using the NICHD Observational Record of the Caregiving Environment (ORCE). Interactions are coded on 4 to 5-point scales including: (1) sensitivity/responsiveness to non-distress, (2) intrusiveness, (3) detachment/disengagement, (4) positive regard for the child, (5) sensitivity/responsiveness to distress, and child distress.

SECONDARY OUTCOMES:
Change in maternal reflective functioning | baseline, 6 months
  The Parental Reflective Functioning Questionnaire (PRFQ-1) measures mothers' reflective functioning and contains 39 statements with instructions to rate each one according to a 7-point Likert scale from 1 ("strongly disagree") to 7 ("strongly agree"), with 4 representing "neutral" or "undecided." The items were formulated to be scored according to three sub-scales: (a) one with high scores representing increased reflective functioning (eg. "My child and I can feel differently about the same thing."), (b) one with low scores representing increased reflective functioning (eg. "My child knows when I am having a bad day and does things to make it worse."), and (c) one with middle, or neutral, scores representing increased reflective functioning and scores at either extreme representing decreased reflective functioning (eg. "When I get angry with my child, I always know the reason why.")

CONTACTS AND LOCATIONS:
Overall Officials: Barry Zuckerman, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No